CLINICAL TRIAL: NCT03705728
Title: Impact of the Automated Administration of Intravenous Anesthesia Compared to Inhalatory Anesthesia on the Speed of Emergence and the Occurrence of Postoperative Delirium
Brief Title: Automated Administration of Intravenous Compared With Inhalatory Anesthesia on the Occurrence of Postoperative Delirium
Acronym: AG-DPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Clinical, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG-DPO
Record Dates: First submitted 2018-10-02; First posted 2018-10-15 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Delirium; Elderly Patient; General Anesthetic Drug Adverse Reaction
Keywords: anesthesia, general; postoperative delirium; postoperative nausea and vomiting; elderly; total intravenous anesthesia; closed-loop anesthesia; EEG monitoring; propofol; remifentanil; sevoflurane
MeSH Terms: conditions — Emergence Delirium; Postoperative Nausea and Vomiting | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: prospective randomized
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous group (Experimental): Propofol & remifentanil administration using the closed-loop controller with the "Easy-TIVA" platfrom.
  Interventions: Drug: Propofol; Drug: Remifentanil automatic
- volatile anesthesia group (Active Comparator): Sevoflurane will be administered manually according to the BIS values. Remifentanil will be administered manually using a Target Controlled Infusion pump using the Minto model.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil manual

INTERVENTIONS:
Drug: Propofol — Propofol will be automatically administered according to the "EasyTIVA" device algorythm to maintain the BIS value within the 40-60 interval
  Arms: Intravenous group
Drug: Sevoflurane — Sevoflurane will be manually administered to maintain the BIS value within the 40-60 interval
  Arms: volatile anesthesia group
Drug: Remifentanil automatic — Remifentanil will be automatically administered according to the "EasyTIVA" device algorythm to maintain the BIS value within the 40-60 interval
  Arms: Intravenous group
Drug: Remifentanil manual — Remifentanil will be manually administered to maintain the BIS value within the 40-60 interval
  Arms: volatile anesthesia group

SUMMARY:
The intravenous administration of anesthetic agents by a controller automatically-guided by an index of cerebral activity (i.e. the bispectral index) decreases the incidence of postoperative delirium, compared with an inhalational anesthesia.

DETAILED DESCRIPTION:
Scientific background Postoperative delirium (POD) is a common complication occurring in 5 to 50 % of elderly patients following an operation. Delirium is a serious complication leading to many medical as well as social and economical consequences. Several studies suggest that, both, the choice of anesthetic agents and the conduction of anesthesia might decrease the incidence of POD.

Objectives Study goal and primary aim: the intravenous administration of anesthetic agents by a controller automatically-guided by an index of cerebral activity (i.e. the bispectral index) decreases the incidence of POD, compared with an inhalational anesthesia.

The primary aim of the present study (i.e. incidence of POD) will be assessed by the Nursing Delirium Screening Scale (NDSS).

Secondary aims:

Secondary aim 1: Assessment of a potential difference on the incidence of PONV between the 2 groups of patients (i.e. intravenous vs. inhaled) by comparison of the number of episodes of nausea and vomiting and the need to treat this complications, between both groups.

Secondary aim 2: study if the difference of in the impairment of cognitive function might be correlated either with the type of drugs used to conduct anesthesia or with the control the index of cerebral activity (i.e. the BIS). The respective influences of the control of the index of cerebral activity (i.e. the BIS) and of the anesthetic drugs on the occurrence of postoperative cognitive dysfunctions (POCD) will be assessed by comparing cognitive function tests on matched groups on the percentage of time spent in different ranges of values of the cortical index Population of patients Patients of 60 years old or more, having given their written informed consent and who should undergo a surgical procedure of at least one hour.

Inclusion criterion

Patients will be included in the study if:

* They are 60 years old or older,
* They have given their written informed consent,
* They have to undergo a surgical procedure of one hour or longer. Non-inclusion criterion

Following patients will non be eligible for the current study:

* Pregnant women,
* Patients presenting a contra-indication to the monitoring of cerebral activity (i.e. intracranial surgery, neuroleptic or anti epileptic medications, pace maker),
* Patients presenting any allergy to propofol and or remifentanil,
* Patients under guardianship. Experimental protocol Information and inclusion of patients during the preoperative anesthetic assessment consultation First assessment of the NDSS at patient arrival in the operating room Randomization prior to the induction on the anesthesia Second NDSS just before patient leaving of PACU Recording of all PONV event as well as any administration of anti emetic drug

Number of subjects: 1000 Number of center: 4 Duration of the research: 36 months

Statistical Analysis: Sequential group analysis. The preoperative and postoperative NDSS test will be analyzed with an ANOVA for repeated-measure and multiple-comparison.

The main criterion will be analyzed with a Kaplan-Meier survival analysis on the global data and with a Cox regression that will take into account the qualitative factors represented by the type of anesthesia

Description of the Nursing Delirium Screening Scale (NDSS) that is a validated scale to assess POD at the bedside.

Five areas are assessed: disorientation, inappropriate behavior, inappropriate communication, illusions or hallucinations, and psychomotor retardation Description A screening tool designed for nurses to use at the end of their shift to identify patients with delirium, derived from the Confusion Rating Scale (CRS). Raters reference behaviors that they have witnessed in the patient or that the patient'snurse has witnessed during their shift to score the NDSS.

The NDSS can be rated one or more times daily.

Scoring information Each feature is scored on 0-2 based on severity, with 0=absent, 1=mild, and 2=severe.

Positive NDSS is score ≥ 2, maximum total score is 10.

ELIGIBILITY:
Inclusion Criteria:

* age > 59 year
* Informed written consent before enrolment;
* Procedure duration > 60 min.
* Speaking French
* Possible contact one-month following surgery

Exclusion Criteria:

* Contraindication of brain monitoring (intracranial surgery), pace-maker.
* Propofol or remifentanil allergy.
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Nurse Delirium Screening Scale in the early postoperative period between intravenous vs halogenated general anesthesia | Measure of the Nurse Delirium Screening Scale, up to an estimated maximum of 3 hours postoperatively
  occurrence of POD as measured by the Nursing Delirium Screening Scale
  The Nursing Delirium Scale
  Symptom Symptom rating Disorientation 0 points 1 point 2 points Inappropriate behavior 0 points 1 point 2 points Inappropriate communication 0 points 1 point 2 points Illusion/hallucination 0 points 1 point 2 points Psychomotot retardation 0 points 1 point 2 points
  Total score ≤ 2 points > 2 points Delirium No Yes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Clinical, Soyaux, Charente, France

REFERENCES:
- [Background] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Background] Besch G, Liu N, Samain E, Pericard C, Boichut N, Mercier M, Chazot T, Pili-Floury S. Occurrence of and risk factors for electroencephalogram burst suppression during propofol-remifentanil anaesthesia. Br J Anaesth. 2011 Nov;107(5):749-56. doi: 10.1093/bja/aer235. Epub 2011 Aug 8. PMID 21828343
- [Background] Liu N, Lory C, Assenzo V, Cocard V, Chazot T, Le Guen M, Sessler DI, Journois D, Fischler M. Feasibility of closed-loop co-administration of propofol and remifentanil guided by the bispectral index in obese patients: a prospective cohort comparison. Br J Anaesth. 2015 Apr;114(4):605-14. doi: 10.1093/bja/aeu401. Epub 2014 Dec 10. PMID 25500680
- [Background] Orliaguet GA, Benabbes Lambert F, Chazot T, Glasman P, Fischler M, Liu N. Feasibility of closed-loop titration of propofol and remifentanil guided by the bispectral monitor in pediatric and adolescent patients: a prospective randomized study. Anesthesiology. 2015 Apr;122(4):759-67. doi: 10.1097/ALN.0000000000000577. PMID 25545655
- [Background] Liu N, Chazot T, Trillat B, Michel-Cherqui M, Marandon JY, Law-Koune JD, Rives B, Fischler M; Foch Lung Transplant Group. Closed-loop control of consciousness during lung transplantation: an observational study. J Cardiothorac Vasc Anesth. 2008 Aug;22(4):611-5. doi: 10.1053/j.jvca.2008.04.022. Epub 2008 Jun 25. PMID 18662642